CLINICAL TRIAL: NCT00981227
Title: Efficacy and Safety of Eslicarbazepine Acetate (BIA 2093) as Therapy for Patients With Post-herpetic Neuralgia: a Double-blind, Double-dummy, Randomised, Placebo-controlled, Parallel-group, Multicentre Clinical Trial
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate as Therapy for Patients With Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-207
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Postherpetic Neuralgia
Keywords: pain herpetic neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- ESL 400 mg twice-daily (Experimental): ESL 400 mg twice-daily
  Interventions: Drug: Eslicarbazepine acetate
- ESL 800 mg once-daily (Experimental): ESL 800 mg once-daily
  Interventions: Drug: Eslicarbazepine acetate
- ESL 600 mg twice daily (Experimental): ESL 600 mg twice daily
  Interventions: Drug: Eslicarbazepine acetate
- ESL 1200 mg once daily (Experimental): ESL 1200 mg once daily
  Interventions: Drug: Eslicarbazepine acetate
- ESL 800 mg twice daily (Experimental): ESL 800 mg twice daily
  Interventions: Drug: Eslicarbazepine acetate
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine acetate — Scored tablets
  Other Names: Zebinix
  Arms: ESL 1200 mg once daily; ESL 400 mg twice-daily; ESL 600 mg twice daily; ESL 800 mg once-daily; ESL 800 mg twice daily
Drug: Placebo — oral route
  Arms: placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of eslicarbazepine acetate (ESL) as therapy for patients with post-herpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Men and women aged 18 years or older
* Previous diagnosis of herpes zoster
* Diagnosis of postherpetic neuralgia and neuropathic pain present for more than 3 months after healing of the herpes zoster skin rash
* Cooperation and willingness to complete all aspects of the study
* Completion of at least 4 daily diaries during the week preceding randomisation
* A minimum average daily pain score of 4 on the NRPS in the last 4 diary entries before randomisation.

Exclusion Criteria:

* Pain of other origin that might confound the assessment of neuropathic pain of postherpetic origin
* Active herpes zoster lesion or dermatitis of any origin at the affected site
* Subjects who had neurological ablation by block or neurosurgical intervention for control of pain
* Significant or unstable medical or psychiatric disorders
* Drug or alcohol abuse in the preceding 2 years
* Severe renal function impairment, as shown by calculated creatinine clearance values < 30 mL/min at screening
* Relevant clinical laboratory abnormalities (e.g., Na+ <130 mmol/L, alanine (ALT) or aspartate (AST) transaminases >2.0 times the upper limit of the normal, white blood cell count (WBC) <2,500 cells/mm3)
* Previous participation in any study with eslicarbazepine acetate
* Pregnancy or breast feeding
* History of hypersensitivity to the investigational products or to drugs with a similar chemical structure
* History of non-compliance
* Likelihood of requiring treatment during the study period with drugs or other interventions not permitted by the clinical study protocol
* Participation in a clinical study within 3 months prior to screening
* Any clinical significant concomitant condition which might influence the assessments or conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 06 November 2007; Date last subject completed: 19 January 2009.
  Number of subjects:
  Planned: 540 subjects (90 in each of the 6 treatment groups). Randomised and treated: 567. Analysed for efficacy (per-protocol): 396 Analysed for safety: 567.
Pre-assignment Details: An up to 2-week baseline was followed by a 1-week titration period, an 8-week maintenance period, and a 2-week safety follow-up period. If subjects had a creatinine clearance between 30 and 60 mL/min, they received half of the assigned dose, and subjects with a creatinine clearance below 30 mL/min were not enrolled in this study.
Groups:
- ESL 1200 mg Once Daily: ESL 1200 mg once daily
  Eslicarbazepine acetate : Scored tablets
- ESL 400 mg Twice-daily: ESL 400 mg twice-daily
  Eslicarbazepine acetate : Scored tablets
- ESL 600 mg Twice Daily: ESL 600 mg twice daily
  Eslicarbazepine acetate : Scored tablets
- ESL 800 mg Once-daily: ESL 800 mg once-daily
  Eslicarbazepine acetate : Scored tablets
- ESL 800 mg Twice Daily: ESL 800 mg twice daily
  Eslicarbazepine acetate : Scored tablets
- Placebo: placebo
  Placebo : oral route
Period: Overall Study
Arm/Group | ESL 1200 mg Once Daily | ESL 400 mg Twice-daily | ESL 600 mg Twice Daily | ESL 800 mg Once-daily | ESL 800 mg Twice Daily | Placebo
Started | 102 | 94 | 94 | 94 | 90 | 93
Randomized | 102 | 94 | 94 | 94 | 90 | 93
Safety Population | 102 | 94 | 94 | 94 | 90 | 93
Per-Protocol | 69 | 72 | 67 | 68 | 50 | 70
Completed | 80 | 75 | 73 | 73 | 60 | 75
Not Completed | 22 | 19 | 21 | 21 | 30 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESL 1200 mg Once Daily | ESL 400 mg Twice-daily | ESL 600 mg Twice Daily | ESL 800 mg Once-daily | ESL 800 mg Twice Daily | Placebo | Total
Number analyzed (Participants) | 102 | 94 | 94 | 94 | 90 | 93 | 567
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 36 | 35 | 37 | 30 | 38 | 210
  >=65 years | 68 | 58 | 59 | 57 | 60 | 55 | 357
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 55 | 57 | 52 | 64 | 44 | 341
  Male | 33 | 39 | 37 | 42 | 26 | 49 | 226

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Pain (NRPS) From Baseline to Endpoint in Mean Pain
Description: The primary efficacy variable will be based upon an 11-point (0-10) Numeric Rating Pain Scale (NRPS), where 0 = no pain and 10 = worst possible pain, to be recorded in a patient's diary upon awakening each morning. This score should reflect the patient's mean pain over the previous 24 hours.
  Please note that the change from baseline to endpoint in mean pain, i.e. the difference between endpoint mean pain and baseline mean pain, which are defined as follows:
  * Baseline mean pain is defined as the mean of the last four available ratings of average daily pain (NRPS) in the patient diary performed in the last 7 days before randomisation.
  * Endpoint mean pain is defined as the mean of the last four available ratings of average daily pain in the patient diary in the last 7 days of the treatment period.
Time Frame: baseline and 13 weeks
Measure: Least Squares Mean (Standard Error); unit: Points
Groups:
- ESL 1200 mg Once Daily; ESL 400 mg Twice-daily; ESL 600 mg Twice Daily; ESL 800 mg Once-daily; ESL 800 mg Twice Daily; Placebo: total daily dose;oral route
Arm/Group | ESL 1200 mg Once Daily | ESL 400 mg Twice-daily | ESL 600 mg Twice Daily | ESL 800 mg Once-daily | ESL 800 mg Twice Daily | Placebo
Number analyzed (Participants) | 102 | 94 | 94 | 92 | 87 | 92
Points | -1.9447 (0.2088) | -1.9786 (0.2178) | -1.6798 (0.2179) | -1.6633 (0.2217) | -2.0834 (0.2280) | -1.5441 (0.2197)

2. Other Pre Specified Outcome: Change in Mean Pain (NRPS) From Baseline to Endpoint by Total Daily Dose
Description: Details of neuropathic pain, as recorded in a subject diary, were used for the primary assessment of analgesic efficacy. Subjects assessed their pain using an 11-point (0 "no pain" to 10 "worst possible pain") NRPS upon awakening each morning and recorded the results in the subject diary. This score reflected the subject's mean pain over the previous 24 hours. Subjects were trained how to record their pain reliably. Investigators were trained in the subject's NRPS use during site initiation visits and at the investigators' meeting.
Time Frame: baseline and 13 weeks
Measure: Least Squares Mean (Standard Error); unit: Points
Groups:
- ESL 1200 mg/Day; ESL 1600 mg/Day; ESL 800 mg/Day: total daily dose;oral route
Arm/Group | Placebo | ESL 1200 mg/Day | ESL 1600 mg/Day | ESL 800 mg/Day
Number analyzed (Participants) | 92 | 196 | 87 | 186
Points | -1.5448 (0.2196) | -1.8183 (0.1512) | -2.0854 (0.2279) | -1.8236 (0.1565)

ADVERSE EVENTS:
Time Frame: All TEAEs, i.e. those AEs starting after the first dose intake until 2 days after the last dose,have been summarized
Arm/Group | ESL 1200 mg Once Daily | ESL 400 mg Twice-daily | ESL 600 mg Twice Daily | ESL 800 mg Once-daily | ESL 800 mg Twice Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 1/102 | 4/94 | 4/94 | 2/94 | 1/90 | 0/93
Other Adverse Events (participants affected / at risk) | 48/102 | 41/94 | 42/94 | 46/94 | 49/90 | 29/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESL 1200 mg Once Daily (N=102) | ESL 400 mg Twice-daily (N=94) | ESL 600 mg Twice Daily (N=94) | ESL 800 mg Once-daily (N=94) | ESL 800 mg Twice Daily (N=90) | Placebo (N=93)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESL 1200 mg Once Daily (N=102) | ESL 400 mg Twice-daily (N=94) | ESL 600 mg Twice Daily (N=94) | ESL 800 mg Once-daily (N=94) | ESL 800 mg Twice Daily (N=90) | Placebo (N=93)
Dizziness (Nervous system disorders) | 9 (9) | 4 (4) | 8 (8) | 5 (5) | 11 (11) | 2 (2)
Somnolence (Nervous system disorders) | 6 (6) | 3 (3) | 2 (2) | 1 (1) | 10 (10) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 3 (3) | 5 (5) | 3 (3) | 8 (8) | 4 (4)
Nausea (Gastrointestinal disorders) | 11 (11) | 3 (3) | 6 (6) | 3 (3) | 8 (8) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4) | 7 (7) | 4 (4) | 6 (6) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 1 (1)
Asthenia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Fatigue (General disorders) | 4 (4) | 6 (6) | 4 (4) | 4 (4) | 3 (3) | 1 (1)
GGT increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other